CLINICAL TRIAL: NCT03998020
Title: Constitution of a Clinical, Neurophysiological and Biological Cohort for Chronic Sleep Disorders Responsible of Hypersomnolence
Acronym: Somnobank
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U1061 Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9895
Record Dates: First submitted 2018-09-10; First posted 2019-06-25 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Somnolence Disorder, Excessive
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Intervention = Blood withdrawal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic sleep disorders (Other): Subjects with chronic sleep disorders responsible of hypersomnolence measured by a scale of severity of sleep disorder, and blood parameters (blood sample)
  Interventions: Other: scale of severity; Genetic: blood sample

INTERVENTIONS:
Other: scale of severity — assessment of the severity of the sleep disorders by scale
Genetic: blood sample — Genetical study, serum and sample

SUMMARY:
Chronic sleep disorders result from multiple pathophysiological mechanisms and are often associated with severe hypersomnolence, responsible for major disability. Hypersomnolence may be secondary to sleep disturbances at night by sleep fragmentation, both overall in restless leg syndrome (RLS) or specific to slow or paradoxical sleep in parasomnias (sleepwalking, sleep behavior disorder). paradoxical). Attention-Deficit / Hyperactivity Disorder (ADHD) is another cause of secondary hypersomnolence, unsolved pathophysiology, leading to a major disturbance of alertness. More rarely, hypersomnolence may be primary (central hypersomnia), representing then the most severe form existing in humans. The best-known central hypersomnia is narcolepsy type 1 (NT1), affecting 0.02% of the population. It is thanks to the existence of well-characterized clinical, biological and neuropathological patients that its pathophysiology is better understood. It is due to a selective loss of hypothalamic neurons secreting orexin / hypocretin, in connection with a probable autoimmune process, in genetically predisposed subjects. Narcolepsy type 2 (NT2), idiopathic hypersomnia (HI) and Kleine-Levin syndrome (SKL), are rarer forms of central hypersomnia, the pathophysiology of which is still unknown, due to the small number of patients studied.

DETAILED DESCRIPTION:
Chronic sleep disorders result from multiple pathophysiological mechanisms and are often associated with severe hypersomnolence, responsible for major disability. Hypersomnolence may be secondary to sleep disturbances at night by sleep fragmentation, both overall in restless leg syndrome (RLS) or specific to slow or paradoxical sleep in parasomnias (sleepwalking, sleep behavior disorder). paradoxical). Attention-Deficit / Hyperactivity Disorder (ADHD) is another cause of secondary hypersomnolence, unsolved pathophysiology, leading to a major disturbance of alertness. More rarely, hypersomnolence may be primary (central hypersomnia), representing then the most severe form existing in humans. The best-known central hypersomnia is narcolepsy type 1 (NT1), affecting 0.02% of the population. It is thanks to the existence of well-characterized clinical, biological and neuropathological patients that its pathophysiology is better understood. It is due to a selective loss of hypothalamic neurons secreting orexin / hypocretin, in connection with a probable autoimmune process, in genetically predisposed subjects. Narcolepsy type 2 (NT2), idiopathic hypersomnia (HI) and Kleine-Levin syndrome (SKL), are rarer forms of central hypersomnia, the pathophysiology of which is still unknown, due to the small number of patients studied.

Chronic sleep disorders result from multiple pathophysiological mechanisms and the constitution of a clinical, neurophysiological and biological cohort, monocentric. Patients (minors or adults) suffering from chronic sleep disorders responsible for hypersomnolence will be recruited, followed by the Sleep Disorders Unit (UTSE) and the National Reference Center for Rare Hypersomnia (CNRH) in Montpellier. The number of topics to include depends on feasibility criteria including the rarity of certain sleep disorders and recruitment opportunities. At a minimum, 150 subjects per group will be recruited according to the following ratio: NT1 (33%), other central hypersomnias (NT2, HI, SKL, 33%), and hypersomnolence secondary to a neurological sleep or vigilance disorder (ADHD, RLS, parasomnias, 33%). A match on age and sex will be considered

ELIGIBILITY:
Inclusion Criteria:

* Have a complaint of chronic hypersomnolence on questioning, identified by a sleep specialist and requiring objective explorations in the Centre de Hypersomnias Rares, with or without a diagnosis of chronic sleep disorder according to the International Classification scale in force at the time of diagnosis
* can be treated or not for chronic sleep disorder.
* speak and understand french
* should have a social security system
* should not have infectious or inflammatory pathology

Exclusion Criteria:

* be private of liberty
* live in medical institution
* be a major protected by law
* not have social security system
* refuse to participate in protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2030-06-16 (Estimated); Study Completion 2033-06-16 (Estimated)

PRIMARY OUTCOMES:
Severity of somnolence | Inclusion
  evaluation with sleep latency test, validated questionnaires

SECONDARY OUTCOMES:
level of somnolence | 12 months maximum
  Physicians Global Assessment to measure the evolution of somnolence

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No